CLINICAL TRIAL: NCT02248064
Title: The Assessment of Intelligent Oxygen Therapy (iO2t) in Patients With Chronic Obstructive Pulmonary Disease (COPD) and Idiopathic Pulmonary Fibrosis (IPF)
Brief Title: Auto-titrating Oxygen in Chronic Respiratory Failure
Acronym: ASI1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: 14IC1995
Record Dates: First submitted 2014-09-12; First posted 2014-09-25 (Estimated); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Chronic Obstructive Pulmonary Disease; Idiopathic Pulmonary Fibrosis
Keywords: Chronic obstructive pulmonary disease; Long term oxygen therapy; Auto-titrating oxygen system; Intelligent oxygen therapy; Idiopathic pulmonary fibrosis
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Idiopathic Pulmonary Fibrosis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Fixed flow oxygen COPD (No Intervention): The 6MWT will done on the patients usual fixed flow ambulatory oxygen in this arm.
- Auto-titrating arm COPD (Experimental): The 6MWT will done using the auto-titrating oxygen system in this arm of the study
  Interventions: Device: Auto-titrating oxygen system
- Fixed flow oxygen Pulmonary Fibrosis (IPF) (No Intervention): The 6MWT will done using the auto-titrating oxygen system in this arm of the study
- Auto-titrating arm Pulmonary Fibrosis (IPF) (Experimental): The 6MWT will done using the auto-titrating oxygen system in this arm of the study
  Interventions: Device: Auto-titrating oxygen system

INTERVENTIONS:
Device: Auto-titrating oxygen system — The auto-titrating oxygen system contains a number of components working together to produce variable oxygen flow. An oximeter measures the oxygen saturation of a patient and via Bluetooth this is relayed to a control centre in a mobile phone. This in turn regulates a flow meter which adjust oxygen flow.
  Other Names: Intelligent oxygen therapy; iO2t
  Arms: Auto-titrating arm COPD; Auto-titrating arm Pulmonary Fibrosis (IPF)

SUMMARY:
Long term oxygen therapy (LTOT) increases the life span of patients with chronic obstructive pulmonary disease who have low oxygen levels. However, even when on oxygen therapy at home, from time to time patients still have low oxygen levels especially when walking which can be harmful.

The investigators have designed a new system of delivering oxygen to overcome the above problem. The system measures the oxygen saturations of a patient and subsequently adjust the flow of oxygen to meet a pre-set oxygen saturation target.

Hypothesis: the investigators intelligent oxygen therapy system is better at reducing low levels of oxygen during a 6 minute walk than usual ambulatory oxygen for patients with chronic obstructive pulmonary disease and idiopathic pulmonary fibrosis.

DETAILED DESCRIPTION:
For patients with chronic obstructive pulmonary disease (COPD) and idiopathic pulmonary fibrosis (IPF), disease progression leads to hypoxic respiratory failure necessitating the use of long-term oxygen therapy (LTOT). However a number of studies have shown that despite being on LTOT at home many patients with COPD still experience episodes of intermittent hypoxia (reduction in oxygen saturation <90%). These episodes occur during rest, sleep, talking, walking and sleep. These episodes of intermittent hypoxia can be harmful as they can lead to the development of ischaemic heart disease, induce pulmonary hypertension and affect brain function.

In order to reduce these episodes of intermittent hypoxia, the investigators have designed an auto-titrating, closed-loop oxygen system which automatically adjust the flow of oxygen to match a given oxygen saturation target. This allows individualisation and optimisation of oxygen therapy for every patient.

Mechanism of action:

A pulse oximeter is attached to the ear or finger of a patient. This send the oxygen saturation reading to a control centre (located in a mobile phone). The control centre is pre-programmed to maintain a set oxygen saturation target. The control centre outputs a signal to a flow meter which regulated the outflow of oxygen.

In this study, the investigators will recruit patients with COPD on LTOT and patients with IPF on LTOT or ambulatory oxygen to undergo three 6 minute walk tests (6MWT). The first will be on air (practice walk), the second will be on their usual ambulatory oxygen and the third on the auto-titrating oxygen system. The order of the second and third walks be randomly selected. The patient will be blinded as to which type of oxygen they will be receiving in the second and third walk.

Hypothesis: the investigators iO2t system is better at preventing and treating oxygen desaturations that occur during a 6MWT than usual fixed flow ambulatory oxygen therapy

ELIGIBILITY:
Inclusion Criteria:

* COPD and on LTOT
* IPF on LTOT or ambulatory oxgen

Exclusion Criteria:

* Unable to mobilise for a 6 minute walk test
* Unable to consent to study,
* Partial pressure of oxygen < 6.0 kilopascals (kPa) or Partial pressure of carbon dioxide > 8kilopascals on air,
* Exacerbation of the underlying lung disease in the previous 4 weeks
* Unstable cardiovascular disease (e.g. arrhythmia, hypertension/hypotension or angina)
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2014-07; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
The percentage of time spent with oxygen saturation below 90% | Assessed at the completion of the 6 minute walk test/s
  The participants complete three 6 minute walk tests. There is continuous oxygen saturation monitoring throughout the walk. At the completion of the walk, the percentage of time spent below an oxgen saturation of 90% is calculated

SECONDARY OUTCOMES:
Total distance walked | Assessed at the completion of the 6 minute walk test
Mean oxygen saturation | Assessed during the 6MWT
Total Volume of oxygen delivered | Assessed at the completion of the 6 minute walk test
  The system records the outflow of oxygen every second. From this data, I can calculate the total volume of oxygen delivered to the patient.

CONTACTS AND LOCATIONS:
Overall Officials: Anita K Simonds, MBBS MD FRCP, Principal Investigator — Royal Brompton & Harefield NHS Foundation Trust
Locations (1):
- Royal Brompton and Harefield NHS Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Moghal, M, Goburdhun, R, Hopkinson, N, Man, W, Morrell, M, Dickinson, R et al. An auto-titrating intelligent oxygen therapy (iO 2 T) system in COPD patients: A randomised cross-over trial. European Respiratory Journal. (2015). 46. OA3281. 10.1183/13993003.congress-2015.OA3281.
- See also: This is completed PhD thesis of M Moghal which includes results to this study Autotitrating oxygen in Chronic Respiratory Failure — https://spiral.imperial.ac.uk/handle/10044/1/59707